CLINICAL TRIAL: NCT02963662
Title: Impact of Gut Hormone and Inflammatory Adipokines in Obese Patients Underwent Bariatric Surgery
Brief Title: Impact of Gut Hormones and Inflammatory Adipokines in Obese Patients Underwent Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gao Zhiguang (Other)
Responsible Party: Sponsor-Investigator, Gao Zhiguang, doctor, First Affiliated Hospital of Jinan University
Organization: First Affiliated Hospital of Jinan University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2014A020212219
Record Dates: First submitted 2016-08-17; First posted 2016-11-15 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Obesity; Chronic Inflammation; Type 2 Diabetes
Keywords: obesity; bariatric surgery; gut hormones; inflammatory adipokine
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Roux-en-Y gastric bypass group (Experimental): The patients undergo Roux-en-Y gastric bypass (RYGB group) following a comprehensive evaluation for the surgical indication
  Interventions: Procedure: laparoscopic Roux-en-Y gastric bypass
- sleeve gastrectomy group (Experimental): The patients undergo sleeve gastrectomy (SG group) following a comprehensive evaluation for the surgical indication
  Interventions: Procedure: laparoscopic sleeve gastrectomy
- Normal BMI group (No Intervention): no intervention

INTERVENTIONS:
Procedure: laparoscopic Roux-en-Y gastric bypass — Laparoscopic Roux-en-Y gastric bypass was one of the interventions pre-specified to be administered to participants. The patients undergo Roux-en-Y gastric bypass (RYGB group) following a comprehensive evaluation for the surgical indication
  Arms: Roux-en-Y gastric bypass group
Procedure: laparoscopic sleeve gastrectomy — Laparoscopic sleeve gastrectomy was the other intervention pre-specified to be administered to participants. The patients undergo sleeve gastrectomy (SG group) following a comprehensive evaluation for the surgical indication
  Arms: sleeve gastrectomy group

SUMMARY:
Obesity and type 2 diabetes, dyslipidemia and related metabolic disease has become a threat to our national life and health which is showing a trend. Bariatric Surgery had been confirmed definite therapeutic effect to obesity and type 2 diabetes. However, laparoscopic gastric bypass and laparoscopic sleeve gastrectomy have the similar outcome to type 2 diabetes, but the two surgical methods and principles are completely different, which mechanisms are not yet clear. Lots of literature report adipose tissue releases adipokines and inflammatory cytokines induced chronic inflammation and obesity-related complications (insulin resistance and Type 2 diabetes).It is not clear whether to change these gastrointestinal hormones, adipokines and secretion of inflammatory cytokines with the operation, which play a therapeutic effect of obesity-related complications and diabetes. In addition, the investigators are wonder whether gut hormones, adipokines and inflammatory cytokines have some correlation in different severity obese patients,. It is worth to explore that could intestinal hormones, adipokines and inflammatory factors levels guide us to choice the different surgical approach to different severity obese patients. The investigators tried to investigate different surgical methods to alleviate diabetes and other metabolic diseases mechanisms though hormones and inflammatory factors and adipose tissue inflammation level and compare the impact of intestinal hormones and inflammatory adipokines of the two surgical approaches.

ELIGIBILITY:
Inclusion Criteria:

* According to the standard of obesity Obesity Task Force established in 2001, BMI≥28k / m2 with obesity-related metabolic diseases in patients, or BMI≥35kg / m2 in patients with severe obesity were selected.
* The age of 14-65 years.
* Self-capacity, non-drug dependence, psychological illness.
* Not prompted stomach ulcers, erosions, tumors, polyps, atrophic gastritis and other stomach diseases in the preoperative endoscopy.
* No history of stomach and abdominal surgery.
* Case Source: First Affiliated Hospital of Jinan University, by the same team of doctors performed the surgical procedure.

Exclusion Criteria:

* Whom did not follow the inclusion criteria

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-10; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
The levels of Ghrelin, Peptide YY,Glucagon,Gastric Inhibitory Peptide ,and GLP2 in the fasting state at preoperation in patients with BMI ≥35 kg/m2 or BMI ≥28 kg/m2 and T2D or metabolic syndrome. | within 4 hours
  Units of gut hormones include Ghrelin in pg/m，Peptide YY in pg/ml，Glucagon in pg/ml，Gastric Inhibitory Peptide in pg/ml, GLP2 in pg/ml. Enzyme-Linked Immunosorbent Assay to measure the levels of these gut hormones
The levels of Insulin in the fasting state at preoperation in patients with BMI ≥35 kg/m2 or BMI ≥28 kg/m2 and T2D or metabolic syndrome. | within 4 hours
  The unit of Insulin is ulu/L.Enzyme-Linked Immunosorbent Assay to measure the levels of Insulin
The levels of Leptin in the fasting state at preoperation in patients with BMI ≥35 kg/m2 or BMI ≥28 kg/m2 and T2D or metabolic syndrome. | within 4 hours
  The unit of Leptin is ng/ml.Enzyme-Linked Immunosorbent Assay to measure the levels of Leptin
The levels of GLP1 in the fasting state at preoperation in patients with BMI ≥35 kg/m2 or BMI ≥28 kg/m2 and T2D or metabolic syndrome. | within 4 hours
  The unit of GLP1 is pmol/L.Enzyme-Linked Immunosorbent Assay to measure the levels of GLP1
The levels of adipokines and inflammatory cytokines in the fasting state at preoperation in patients with BMI ≥35 kg/m2 or BMI ≥28 kg/m2 and T2D or metabolic syndrome. | within 4 hours
  Units of adipokines and inflammatory cytokines include Adiponectin in pg/ml, Interleukin 1βin pg/ml , Interleukin 6 in pg/ml, Interleukin 18 in pg/ml, Lipopolysaccharide in pg/ml, NLRP3 in pg/ml, TLR4 in pg/ml, TNF-α in pg/ml.Enzyme-Linked Immunosorbent Assay to measure the levels of adipokines and inflammatory cytokines

SECONDARY OUTCOMES:
The gut hormone levels in the fasting state at 1 month, 3 months, 6 months and 12 months after surgery | 12 months
  "surgery"means laparoscopic gastric bypass or laparoscopic sleeve gastrectomy. Units of gut hormones include Ghrelin in pg/m，Peptide YY in pg/ml，Glucagon in pg/ml，Gastric Inhibitory Peptide in pg/ml, GLP2 in pg/ml.Enzyme-Linked Immunosorbent Assay to measure the levels of these gut hormones
The Insulin levels in the fasting state at 1 month, 3 months, 6 months and 12 months after surgery | 12 months
  The unit of Insulin is ulu/L.Enzyme-Linked Immunosorbent Assay to measure the levels of Insulin.
The Leptin levels in the fasting state at 1 month, 3 months, 6 months and 12 months after surgery | 12 months
  The unit of Leptin is ng/ml.Enzyme-Linked Immunosorbent Assay to measure the levels of Leptin
The GLP1 levels in the fasting state at 1 month, 3 months, 6 months and 12 months after surgery | 12 months
  The unit of GLP1 is pmol/L.Enzyme-Linked Immunosorbent Assay to measure the levels of GLP1
The adipokines and inflammatory cytokines levels in the fasting state at 1 month, 3 months, 6 months and 12 months after surgery | 12 months
  Effect of laparoscopic gastric bypass or laparoscopic sleeve gastrectomy on preoperative and postoperative adipokines and inflammatory cytokines.Units of them include Adiponectin in pg/ml, Interleukin 1βin pg/ml , Interleukin 6 in pg/ml, Interleukin 18 in pg/ml, Lipopolysaccharide in pg/ml, NLRP3 in pg/ml, TLR4 in pg/ml, TNF-α in pg/ml.Enzyme-Linked Immunosorbent Assay to measure the levels of adipokines and inflammatory cytokines.

CONTACTS AND LOCATIONS:
Overall Officials: Jingge Yang, MD,PhD, Principal Investigator — First Affiliated Hospital of Jinan University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yang J, Gao Z, Williams DB, Wang C, Lee S, Zhou X, Qiu P. Effect of laparoscopic Roux-en-Y gastric bypass versus laparoscopic sleeve gastrectomy on fasting gastrointestinal and pancreatic peptide hormones: A prospective nonrandomized trial. Surg Obes Relat Dis. 2018 Oct;14(10):1521-1529. doi: 10.1016/j.soard.2018.06.003. Epub 2018 Jun 14. PMID 30449509